CLINICAL TRIAL: NCT03165734
Title: A Randomized, Controlled Phase 3 Study of Pacritinib Versus Physician's Choice in Patients With Primary Myelofibrosis, Post Polycythemia Vera Myelofibrosis, or Post-Essential Thrombocythemia Myelofibrosis With Severe Thrombocytopenia (Platelet Count <50,000/μL)(PACIFICA)
Brief Title: A Phase 3 Study of Pacritinib in Patients With Primary Myelofibrosis, Post Polycythemia Vera Myelofibrosis, or Post-Essential Thrombocythemia Myelofibrosis
Acronym: PACIFICA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: PSI CRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAC203/PAC303; PAC303 (Other: Sobi, Inc.)
Record Dates: First submitted 2017-05-17; First posted 2017-05-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-10

CONDITIONS: Primary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis
Keywords: myelofibrosis; pacritinib; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis; Ruxolitinib; Bone Marrow Disease; Hematologic Diseases; Blood Platelet Disorders; Hemorrhagic Disorders; Splenomegaly; Anemia; Spleen volume; Spleen
MeSH Terms: conditions — Primary Myelofibrosis; Bone Marrow Diseases; Hematologic Diseases; Blood Platelet Disorders; Hemorrhagic Disorders; Splenomegaly; Anemia | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Adrenal Cortex Hormones; Hydroxyurea; Danazol; ruxolitinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pacritinib 200 mg BID (Experimental): To receive pacritinib 200 mg twice daily (BID) orally, at the same time of day, with or without food
  Interventions: Drug: Pacritinib
- Physician's Choice (P/C) therapy (Active Comparator): The Physician's Choice (P/C) therapy (limited to single drugs from the following list: corticosteroids, hydroxyurea, danazol, or low-dose ruxolitinib). The proposed P/C regimen for a patient must be selected prior to randomization.
  Interventions: Drug: Physician's Choice medications

INTERVENTIONS:
Drug: Pacritinib — Oral administration. Supplied in capsules containing 100 mg (as the free base) in red cap/gray body size 0 opaque hard gelatin capsules. The inactive ingredients are microcrystalline cellulose, magnesium stearate, and polyethylene glycol 8000. Each capsule contains 146 mg of pacritinib citrate, which is equivalent to 100 mg pacritinib free base
  Arms: Pacritinib 200 mg BID
Drug: Physician's Choice medications — Physician's Choice medications will be selected and administered according to the investigator's judgement. Investigators can select individual P/C agents but cannot combine agents or give them sequentially.
  Other Names: corticosteroids; hydroxyurea; danazol; low-dose ruxolitinib
  Arms: Physician's Choice (P/C) therapy

SUMMARY:
This study (study ID PAC203 North America; PAC303 ex-North America) is evaluating 200 mg BID of pacritinib compared to physician's choice (P/C) therapy in patients with MF and severe thrombocytopenia (platelet count <50,000/μL). Approximately 399 patients in total will be enrolled, randomized 2:1 to either pacritinib (approximately 266 patients) or to P/C therapy (approximately 133 patients)

Condition or disease: Primary Myelofibrosis/Post-Polycythemia Vera Myelofibrosis/ Post-essential Thrombocythemia Myelofibrosis

Intervention/treatment: Drug-Pacritinib

DETAILED DESCRIPTION:
The study is a randomized, controlled phase 3 study comparing the efficacy of pacritinib with P/C therapy in patients with PMF, PPV-MF, or PET-MF (Dynamic International Prognostic Scoring System [DIPSS] risk score of Intermediate-1 to High-Risk), who have had had no or limited exposure to any JAK2 inhibitor or are JAK2 inhibitor-naive, and who have severe thrombocytopenia (platelet count <50,000/µL). This study was designed to use the pacritinib 200 mg BID dose, which was determined to be the optimal dose based on dose- and exposure-response analyses conducted using all available data, including the dosing data from the previous portion of this study. Patients will be randomized 2:1 to receive pacritinib 200 mg BID or the P/C therapy (limited to single drugs from the following list: corticosteroids, hydroxyurea, danazol, or low-dose ruxolitinib). The proposed P/C regimen for a patient must be selected prior to randomization. Randomization will be stratified by prior JAK2 inhibitor therapy (yes/no) and P/C therapy selected prior to randomization. Prior JAK2 inhibitor therapy will be defined as any duration of treatment with a JAK2 inhibitor, such as ruxolitinib, fedratinib, or momelotinib. To be eligible, patients are not allowed to have been treated with more than one JAK2 inhibitor. Assigned treatment will continue until the patient experiences progressive disease or intolerable AEs, withdraws consent, or initiates new MF-directed therapy. No study treatment crossover will be allowed at any time. All patients should complete all visit procedures through Week 24, including patients who stop treatment or have protocol-defined progressive disease prior to Week 24, unless the patient withdraws consent for study procedures, dies, undergoes splenic irradiation or splenectomy, initiates any non-protocol-directed anti-MF treatment, or the study is terminated. In addition to the above, patients will be considered to have discontinued treatment if pacritinib or P/C therapy is held for >28 consecutive days due to treatment toxicity, or if treatment is discontinued for lack of efficacy, or at the request of the principal investigator or the patient. Following the Week 24 assessment, patients who are benefiting from therapy will be allowed to continue receiving the assigned treatment (pacritinib or P/C) until the patient experiences progressive disease, intolerable AEs, withdraws consent, or initiates new MF-directed therapy. All randomized patients will be followed for survival for 2.5 years from the date of randomization unless consent for follow-up is withdrawn.

ELIGIBILITY:
Diagnosis and Inclusion Criteria

1. Primary MF, post-polycythemia vera MF, or post-essential thrombocythemia MF (as defined by Tefferi and Vardiman 2008)
2. Platelet count of <50,000/μL at Screening (Day -35 to Day -3)
3. Dynamic International Prognostic Scoring System Intermediate-1, Intermediate-2, or High-Risk (Passamonti et al 2010)
4. Palpable splenomegaly ≥5 cm below the lower costal margin in the midclavicular line as assessed by physical examination
5. TSS of ≥10 on the MPN-SAF TSS 2.0 or a single symptom score of ≥5 or two symptoms of ≥3, including only the symptoms of left upper quadrant pain, bone pain, itching, or night sweats. The TSS criteria need only to be met on a single day.
6. Age ≥18 years
7. Eastern Cooperative Oncology Group performance status 0 to 2
8. Peripheral blast count of <10% throughout the Screening period prior to randomization
9. Absolute neutrophil count of ≥500/µL
10. Left ventricular cardiac ejection fraction of ≥50% by echocardiogram or multigated acquisition scan
11. Adequate liver and renal function, defined by liver transaminases (aspartate aminotransferase [AST]/serum glutamic-oxaloacetic transaminase [SGOT] and alanine aminotransferase [ALT]/serum glutamic pyruvic transaminase [SGPT]) ≤3 × the upper limit of normal (ULN) (AST/ALT ≤5 × ULN if transaminase elevation is related to MF), total bilirubin ≤4 x ULN (in cases where total bilirubin is elevated, direct bilirubin ≤4 × ULN, is required) and creatinine ≤2.5 mg/dL
12. Adequate coagulation defined by prothrombin time/international normalized ratio and partial thromboplastin time ≤1.5 × ULN
13. If fertile, willing to use highly effective birth control methods during the study (see Section 7.1.2.6 for acceptable birth control methods)
14. Willing to undergo and able to tolerate frequent MRI or CT scan assessments during the study
15. Able to understand and willing to complete symptom assessments using a patient-reported outcome instrument
16. Provision of signed informed consent

Exclusion Criteria

1. Life expectancy <6 months
2. Completed allogeneic stem cell transplant or are eligible for and willing to complete other approved available therapy including allogeneic stem cell transplant
3. History of splenectomy or planning to undergo splenectomy
4. Splenic irradiation within the last 6 months
5. Previously treated with pacritinib
6. Treatment with any MF-directed therapy within 14 days prior to treatment Day 1
7. Prior treatment with more than one JAK2 inhibitor
8. Prior treatment with with ruxolitinib, if BOTH of the following conditions are met:

   i. exposure to higher-dose ruxolitinib (>10 mg daily) within 120 days prior to treatment Day 1 AND ii. total duration of treatment with higher-dose ruxolitinib (>10 mg daily) was >90 days, from first to last exposure (i.e., this 90-day period starts on the date of first administration of ruxolitinib at a total daily dose of >10 mg and continues for 90 calendar days, regardless of whether higher-dose ruxolitinib is administered continuously or intermittently).
9. Prior treatment with any JAK2 inhibitor other than ruxolitinib, irrespective of dose, with a duration of >90 days. The 90-day period starts on the date of first administration of JAK2 inhibitor therapy and continues for 90 calendar days, regardless of whether therapy is administered continuously or intermittently.
10. Treatment with an experimental therapy, including MF-directed experimental therapies within 28 days prior to treatment Day 1
11. Systemic treatment with a strong cytochrome P450 3A4 (CYP 3A4) inhibitor or a strong CYP 3A4 inducer within 14 days prior to treatment Day 1. Shorter washout periods may be permitted with approval of the Medical Monitor, provided that the washout period is at least five half-lives of the drug prior to treatment Day 1
12. Significant recent bleeding history defined as National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) grade ≥2 within 3 months prior to treatment Day 1, unless precipitated by an inciting event (eg, surgery, trauma, or injury)
13. Systemic treatment with medications that increase the risk of bleeding, including anticoagulants, antiplatelet agents (except for aspirin dosages of ≤100 mg per day),and daily use of cyclooxygenase-1 (COX-1) inhibiting non-steroidal anti-inflammatory drugs (NSAIDs) within 14 days prior to treatment Day 1. Treatment with systemic anti-vascular endothelial growth factor (anti-VEGF) agents within 28 days prior to treatment Day 1.
14. Systemic treatment with medications that can prolong the QT interval within 14 days prior to treatment Day 1. Shorter washout periods may be permitted with approval of the Medical Monitor, provided that the washout period is at least five half-lives of the drug prior to treatment Day 1
15. Any history of CTCAE grade ≥2 non-dysrhythmia cardiac conditions within 6 months prior to treatment Day 1. Patients with asymptomatic grade 2 non-dysrhythmia cardiovascular conditions may be considered for inclusion, with the approval of the Medical Monitor, if stable and unlikely to affect patient safety.
16. Any history of CTCAE grade ≥2 cardiac dysrhythmias within 6 months prior to treatment Day 1. Patients with non-corrected QT interval CTCAE grade 2 cardiac dysrhythmias may be considered for inclusion, with the approval of the Medical Monitor, if the dysrhythmias are stable, asymptomatic, and unlikely to affect patient safety.
17. QT corrected by the Fridericia method (QTcF) prolongation >450 ms or other factors that increase the risk for QT interval prolongation (eg, hypokalemia [defined as serum potassium <3.0 mEq/L that is persistent and refractory to correction], or history of long QT interval syndrome).
18. New York Heart Association Class II, III, or IV congestive heart failure
19. Any active gastrointestinal or metabolic condition that could interfere with absorption of oral medication
20. Active or uncontrolled inflammatory or chronic functional bowel disorder such as Crohn's Disease, inflammatory bowel disease, chronic diarrhea, or chronic constipation
21. Other malignancy within 3 years prior to treatment Day 1. The following patients may be eligible despite having had a malignancy within the prior 3 years: patients with curatively treated squamous or basal cell carcinoma of the skin; patients with curatively treated non-invasive cancers; patients with organ-confined prostate cancer with prostate specific antigen (PSA) <20 ng/mL and National Comprehensive Cancer Network risk of Very Low, Low, or Favorable Intermediate; and patients with curatively treated non-metastatic prostate cancer with negative PSA.
22. Uncontrolled intercurrent illness, including, but not limited to, ongoing active infection, psychiatric illness, or social situation that, in the judgment of the treating physician, would limit compliance with study requirements
23. Known seropositivity for human immunodeficiency (HIV) virus. For patients in Czech Republic, France and Italy only: testing for HIV is required during Screening.
24. Known active hepatitis A, B, or C virus infection. For patients in Czech Republic, France and Italy only: testing for hepatitis B and C is required during Screening.
25. Women who are pregnant or lactating
26. Concurrent enrollment in another interventional trial
27. Severe thrombocytopenia due to vitamin B12 deficiency, folate deficiency, or viral infection in the opinion of the investigator
28. Known hypersensitivity to pacritinib or any of the following inactive ingredients: microcrystalline cellulose, polyethylene glycol, and magnesium stearate; any contraindication to the "physician's choice" medicinal product selected by the investigator to be used as the comparator or to loperamide or equivalent antidiarrheal medication
29. Persons deprived of their liberty by a judicial or administrative decision
30. Persons subject to legal protection measures or unable to express their consent
31. Temporarily incapacitated persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Spleen volume | From baseline at 24 weeks
  To compare the efficacy of pacritinib with that of physician's choice (P/C) therapy, as assessed by the proportion of patients achieving a ≥35% spleen volume reduction (SVR) as measured by magnetic resonance imaging (MRI, preferred) or computed tomography (CT) scans
Total Symptom Score (TSS) (excluding tiredness) | From baseline at Week 24
  To compare the efficacy of pacritinib compared to P/C therapy, as assessed by the proportion of patients achieving a ≥50% reduction in Total Symptom Score (TSS). The TSS is the sum of the individual symptom scores for tiredness, early satiety, abdominal discomfort, night sweats, pruritus, bone pain, and pain under ribs on the left side. Symptoms are ranked 0 (absent) to 10 (worst imaginable)

SECONDARY OUTCOMES:
Overall Survival (OS) | until 2.5 years after the date of randomization
  To compare the overall survival (OS) of patients treated with pacritinib versus those treated with P/C
Patient Global Impression of Change (PGIC) assessed at Week 24 | End of Week 12 to 2 years following Week 24 visit
  To compare the percentage of patients who self-assess as "very much improved" or "much improved" as measured by the Patient Global Impression of Change (PGIC) in patients treated with pacritinib versus those treated with P/C
To compare the safety of pacritinib versus P/C therapy | Randomization through 30 after last treatment
  Safety will be assessed based on the incidence and severity (according to the Common Terminology Criteria for Adverse Events) of treatment emergent adverse events from the time of randomization until 30 days after completion of treatment with pacritinib and/or physician's choice therapy.

OTHER OUTCOMES:
SVR of ≥35% | Up to 24 Weeks
  Time to achievement of SVR of ≥35%
Best response in SVR | At 24 Weeks
  Best response in SVR by MRI or CT scan
>25% SVR | From baseline and at Week 24
  Proportion of patients achieving >25% SVR
Red blood cell (RBC) | Baseline to End of Treatment
  Achievement of red blood cell (RBC) transfusion independence at Weeks 12 and 24
hemoglobin level | Weeks 12 and 24
  Improvement in hemoglobin level without transfusion at Weeks 12 and 24
platelet count | Weeks 12 and 24
  Improvement in platelet count at Weeks 12 and 24
platelet transfusions | Weeks 12 and 24
  Frequency of platelet transfusions at Weeks 12 and 24
PROMIS | Baseline to Week 24
  Improvement in fatigue as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) v.1.0 - Fatigue from Baseline through Week 24
Leukemia-free survival (LFS) | Baseline to Week 24
  Leukemia-free survival (LFS) of patients treated with pacritinib versus P/C therapy
The percentage of red blood cell transfusion-independent patients achieving a 1 g/dL and a 2 g/dL increase in hemoglobin | Baseline to 24 weeks
  The percentage of red blood cell transfusion-independent patients at baseline achieving a 1 g/dL and a 2 g/dL increase in hemoglobin at week 24
The percentage of platelet transfusion-independent patients with improvement in grade of thrombocytopenia | Baseline to 24 weeks
  The percentage of platelet transfusion-independent patients at baseline with improvement in grade of thrombocytopenia at week 24
The percentage of transfusion-dependent patients achieving transfusion independence and achieving 50% reduction in transfusion rate | Baseline to 24 weeks
  The percentage of transfusion-dependent patients at baseline achieving transfusion independence and achieving 50% reduction in transfusion rate at week 24
Hemoglobin A1c | Baseline to Week 24
  Changes in hemoglobin A1c
mutated allelic burden, gene expression, and pharmacodynamic (PD) biomarkers | Baseline to up to 24 Weeks
  Changes in mutated allelic burden, gene expression, and pharmacodynamic (PD) biomarkers
The proportion of patients who experience a major adverse cardiac event (MACE) | Baseline to up to 24 Weeks
  MACE is a composite endpoint that is considered to occur if any of the following TEAEs occur:
  * cardiovascular death, defined as death due to acute myocardial infarction, sudden cardiac death, death due to heart failure, death due to stroke, death due to cardiovascular procedures, death due to cardiovascular hemorrhage, or death due to peripheral artery disease
  * non-fatal myocardial infarction
  * non-fatal stroke of any classification, including reversible focal neurological defects with imaging evidence of a new cerebral lesion consistent with ischemia or hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Simran Singh, Study Director — Sobi, Inc.
Locations (207):
- United States (42):
  - University of Alabama at Birmingham, (UAB) Hospital, Comprehensive Cancer Center, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Rocky Mountain Cancer Centers (US Oncology/McKesson), Boulder, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - George Washington University-Medical Faculty Associates, Washington D.C., District of Columbia
  - Cleveland Clinic Florida, Weston, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Saint Agnes Hospital, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Regional Cancer Care Associates LLC - CCBD Division, Bethesda, Maryland
  - Maryland Oncology Hematology, PA- Columbia, Columbia, Maryland
  - Michigan Medicine Hematology Clinic-Rogel Cancer Center, Ann Arbor, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Washington University School of Medicine-Siteman Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada- Twain Office, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan -Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Hospital, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - The Sarah Cannon Research Institute-Tennessee Oncology, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Mays Cancer Center, San Antonio, Texas
  - Texas Oncology- San Antonio, San Antonio, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (3):
  - Westmead Hospital, Sydney, New South Wales
  - Alfred Hospital, Malignant Hematology and Stem Cell Transplantation Service, Melbourne, Victoria
  - The Perth Blood Institute, Perth, Western Australia
- Belarus (3):
  - Grodno University Hospital, Grodno
  - Republican Research Center for Radiation Medicine and Human Ecology, Homyel
  - Minsk Scientific and Practical Center of Surgery, Transplantology and Hematology, Minsk
- Bosnia and Herzegovina (2):
  - University Clinical Centre of the Republic of Srpska, Banja Luka
  - University Clinical Center of Sarajevo, Sarajevo
- Brazil (15):
  - Integrare Therapeutics, Fortaleza, Ceará
  - Hospital Sao Rafael, Salvador, Estado de Bahia
  - Clinics Hospital, Federal University of Goias - (UFG), Goiânia, Goiás
  - Cetus Oncology Inc., Belo Horizonte, Minas Gerais
  - Clinical Hospital of the Federal University of Parana (HC - UFPR), Curitiba, Paraná
  - Saint Lucas Hospital of Copacabana, Rio de Janeiro, Rio de Janeiro
  - Humane Clinic / Atena Research Institute, Mossoró, Rio Grande do Norte
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Integrated Oncology Center of Rio Grande do Sul - Mother of God Hospital, Porto Alegre, Rio Grande do Sul
  - Santa Catarina Health Research and Education Center (CEPEN), Florianópolis, Santa Catarina
  - State University of Campinas (UNICAMP) - Hemocenter, Campinas, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Jewish Hospital Albert Einstein, São Paulo, São Paulo
  - Samaritano Hospital, São Paulo, São Paulo
  - Sao Paulo University Clinical Hospital, São Paulo, São Paulo
- Bulgaria (5):
  - University Multiprofile Hospital for Active Treatment "Dr. Georgi Stranski", Pleven
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi", Plovdiv, Plovdiv
  - Multiprofile Hospital for Active Treatment - Sofia, part of Military Medical Academy, Sofia
  - Specialized Hospital for Active Treatment of Hematological Diseases, Sofia
  - Multiprofile Hospital for Active Treatment "Sveta Marina", Varna
- Canada (7):
  - Tom Baker Cancer Center, Internal Medicine/Hematology, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Providence Hematology - Vancouver, Vancouver, British Columbia
  - Eastern Regional Health Authority, St. John's, Newfoundland and Labrador
  - Nova Scotia Health Authority, Centre for Clinical Research, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital; Clinical Research Unit, Montreal, Quebec
- Czechia (4):
  - University Hospital Brno, Brno
  - University Hospital Olomouc, Olomouc
  - University Hospital Plzen, Pilsen
  - University Hospital Kralovske Vinohrady, Clinic of Internal Hematology, Prague
- France (7):
  - CHU Hôpital Amiens Sud, Amiens, France
  - CHU de Nimes - Hopital Universitaire Caremeau, Nîmes, France
  - La Conception Hospital, Marseille
  - Hôpital Saint-Louis, Paris
  - CHU Hopitaux de Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - University Hospital Center of Poitiers, Poitiers
- Georgia (5):
  - JSC K. Eristavi National Center For Experimental and Clinical Surgery, Tbilisi
  - LTD M.Zodelava's Hematology Center, Department of Hematology, Tbilisi
  - LTD S.Khechinashvili University Hospital, Tbilisi
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center LTD, Tbilisi
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic LLC, Tbilisi
- Hungary (5):
  - Semmelweis University SE ÁOK I. sz. Belgyógyászati Klinika, Budapest
  - University of Debrecen Clinical Center (Debreceni Egyetem Klinikai Központ), Debrecen
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
  - Szabolcs-Szatmar-Bereg County Hospitals and University Teaching Hospital, Department of Hematology, Nyíregyháza
  - Fejer County St. Gyorgy University Teaching Hospital, Department of Internal Medicine I, Székesfehérvár
- India (13):
  - Gauhati Medical College and Hospital, Guwahati, Assam
  - Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh, Chandigarh
  - Nirmal Hospital Pvt Ltd, Surat, Gujarat
  - Fortis Memorial Research Institute(FMRI), Gurgaon, Haryana
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Shri Ram Cancer Centre, Mahatma Gandhi Medical College & Hospital, Jaipur, Rajasthan
  - Meenakshi Mission Hospital And Research Centre (MMHRC), Madurai, Tamil Nadu
  - Yashoda Hospitals, Hyderabad, Telangana
  - All India Institute of Medical Sciences, Dehradun, Uttarakhand
  - Netaji Subhash Chandra Bose Cancer Research Institute, Kolkata, West Bengal
  - Tata Medical Center, Kolkata, West Bengal
  - St. John's Medical College Hospital, Bengaluru
  - Max Super Speciality Hospital Saket (A Unit of Max Healthcare Institute Limited), Delhi
- Israel (5):
  - Lady Davis Carmel Medical Center, Department of Hematology,, Haifa
  - Hadassah Medical Center, Department of Hematology,, Jerusalem
  - Meir Medical Center, Hematology Institute and Blood Bank, Kfar Saba
  - Rabin Medical Center, Clinic for Myeloproliferative Disorders, Petah Tikva
  - The Tel Aviv Sourasky Medical Center, Department of Internal Medicine, Tel Aviv
- Italy (17):
  - Cancer Institute "Giovanni Paolo II", IRCCS, Bari
  - Polyclinic S. Orsola-Malpighi, Bologna
  - ASST Spedali Civili Brescia, Hematology Unit, Brescia
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Scientific Institute of Romagna for the Study and Treatment of Cancer (IRST), IRCCS, Forlì
  - Maggiore Polyclinic Hospital, Fondazione IRCCS Ca' Granda, Milan
  - ASST Monza - Ospedale San Gerardo, Monza
  - University Hospital "Federico II", Naples
  - University Hospital "Maggiore della Carita" of Novara, Novara
  - United Hospitals Villa Sofia Cervello, Palermo
  - Polyclinic San Matteo, IRCCS, Pavia
  - Hospital "Infermi" of Rimini, Rimini
  - Umberto I Polyclinic of Rome, Rome
  - University Polyclinic Foundation "Agostino Gemelli", Rome
  - City of Health and Science of Turin, Turin
  - Santa Maria della Misericordia University Hospital of Udine, Udine
  - ASST Sette Laghi Hospital, Varese
- Japan (10):
  - University of Yamanashi Hospital, Chūō
  - Kyushu University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Tohoku University Hospital, Miyagi
  - University of Miyazaki Hospital, Miyazaki
  - Juntendo University Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Ehime University Hospital, Tōon
  - Mie University Hospital, Tsu
- Kazakhstan (7):
  - Aktobe Medical Center, Department of Hematology, Aktobe
  - City Clinical Hospital #7, Hematology Department, Almaty
  - Center for Hematology, Astana
  - National Research Oncology, Oncohematology Center, Astana
  - Hematology Center, Karaganda
  - City Oncological Center, Shymkent
  - Center for Hematology, Ust-Kamenogorsk
- Poland (12):
  - University Teaching Hospital in Bialystok, Bialystok
  - University Clinical Center in Gdansk, Gdansk
  - Andrzej Mielecki Independent Public Clinical Hospital of Medical University of Silesia in Katowice, Department of Hematology and Bone Marrow Transplantation, Katowice
  - Pratia Oncology Katowice, Katowice
  - University Hospital in Krakow, Krakow
  - Nicolaus Copernicus Provincial Multispecialty Oncology and Traumatology Center in Lodz, Lodz
  - Independent Public Teaching Hospital No.1 in Lublin, Department of Hematooncology, Bone Marrow Transplantation and Chemotherapy, Lublin
  - Jedrzej Sniadecki Specialist Hospital in Nowy Sacz, Department of Hematology, Nowy Sącz
  - Frederic Chopin Provincial Teaching Hospital No. 1 in Rzeszow, Department of Hematology,, Rzeszów
  - Nasz Lekarz Medical Outpatient Clinics Slawomir Jeka, Torun
  - Institute of Hematology and Transfusion Medicine, Teaching Department of Hematology, Warsaw
  - Jan Mikulicz Radecki University Hospital in Wroclaw, Department and Clinic of Hematology, Blood Neoplasms and Bone Marrow Transplantation, Wroclaw
- Romania (4):
  - Onco Card Srl, Brasov
  - Coltea Clinical Hospital, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - Prof. Dr. Ion Chiricuta" Institute of Oncology, Cluj-Napoca
- Russia (9):
  - City Clinical Hospital #40, Moscow
  - City Clinical Hospital n.a. V.V. Veresaev of the Moscow City Health, Moscow
  - S.P. Botkin City Clinical Hospital, Moscow
  - Clinic UZI 4D, LLC, Pyatigorsk
  - Research Institute of Hematology and Transfusiology, Saint Petersburg
  - S.M. Kirov Military Medical Academy, Department and Clinic for Intermediate-Level Training in Internal Medicine, Hematology Division, Saint Petersburg
  - V.A. Almazov North-West Federal Medical Research Center, Institute of Oncology and Hematology, Scientific Department of Clinical Oncology, Saint Petersburg
  - Bashkiria State Medical University, Department of Internal Medicine, Ufa
  - Volgograd Regional Clinical Oncology Center, Volgograd
- Serbia (2):
  - Clinical Center of Serbia, Clinic of Hematology, Belgrade
  - Clinical Center of Vojvodina, Clinic of Hematology, Novi Sad
- South Korea (6):
  - Severance Hospital, Seoul, South Korea
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, St. Mary's Hospital, Seoul
- Spain (9):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - University Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - University Hospital 12 de Octubre, Department of Hematology, Madrid
  - Morales Meseguer University General Hospital, Department of Hematology and Hemotherapy, Murcia
  - University Clinical Hospital of Salamanca, Department of Hematology, Salamanca
  - University Hospital Virgen del Rocio (HUVR), Seville
  - University Clinical Hospital of Valencia, Department of Hematology and Medical Oncology, Valencia
- Ukraine (8):
  - Cherkasy Regional Oncology Dispensary of Cherkasy Oblast Council, Regional Treatment and Diagnostic Hematology Center, Department of Hematology, Cherkasy
  - City Clinical Hospital #4" under Dnipro City Council, Dnipro
  - Communal Non-profit enterprise "Regional Center of Oncology", Department of Hematology, Kharkiv
  - Kyiv City Clinical Hospital #9, Hematology Department #1, Kyiv
  - Kyiv Regional Oncology Center, Department of Hematology,, Kyiv
  - Limited Liability Company "City Doctor", Kyiv
  - Institute of Blood Pathology and Transfusion Medicine, Department of Hematology, Lviv
  - Poltava M.V. Sklifosovskyi Regional Clinical Hospital under Poltava Regional Council, Department of Hematology, Poltava
- United Kingdom (7):
  - Royal Hallamshire Hospital, Department of Hematology, Sheffield, South Yorkshire
  - Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom
  - Barts Health NHS Trust - The Royal London Hospital, London, United Kingdom
  - Gloucestershire Royal Hospital, Gloucester
  - Guy's and St Thomas' NHS Foundation Trust - Guy's Hospital, London
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital, London
  - Oxford University Hospitals NHS Trust - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerds AT, Savona MR, Scott BL, Talpaz M, Egyed M, Harrison CN, Yacoub A, Vannucchi A, Mead AJ, Kiladjian JJ, O'Sullivan J, Garcia-Gutierrez V, Bose P, Rampal RK, Miller CB, Palmer J, Oh ST, Buckley SA, Mould DR, Ito K, Tyavanagimatt S, Smith JA, Roman-Torres K, Devineni S, Craig AR, Mascarenhas JO. Determining the recommended dose of pacritinib: results from the PAC203 dose-finding trial in advanced myelofibrosis. Blood Adv. 2020 Nov 24;4(22):5825-5835. doi: 10.1182/bloodadvances.2020003314. PMID 33232476